CLINICAL TRIAL: NCT06238973
Title: Evaluation of the Relationship Between the Level of Controlled Hypotension Applied During Rhinoplasty and Septoplasty Surgery and the Incidence of Postoperative Cognitive Dysfunction and Delirium
Brief Title: Controlled Hypotension in Rhinoplasty and Septoplasty: Incidence of Cognitive Dysfunction and Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Selcuk KAYIR, Assossiated Professor, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2023-101
Record Dates: First submitted 2024-01-23; First posted 2024-02-02 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hypotension During Surgery
Keywords: controlled hypotension; nasal surgery; post operative cognitive dysfunction; post operative delirium
MeSH Terms: conditions — Emergence Delirium | interventions — low mobility group protein 160, rat

STUDY DESIGN:
Intervention Model Description: The group to be designated as Group A will aim to maintain an average arterial pressure in the range of 50-57 mmHg. For Group B, the target is to keep the average arterial pressure within the range of 58-65 mmHg.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Low (Active Comparator): Group Low will aim to maintain an average arterial pressure in the range of 50-57 mmHg.
  Interventions: Other: Group Low
- Group Middle (Active Comparator): The target is to keep the average arterial pressure within the range of 58-65 mmHg
  Interventions: Other: Group Middle

INTERVENTIONS:
Other: Group Low — In order to maintain arterial blood pressure within the range of 50-57 mmHg, Sevoflurane at a concentration of 0.5-1 MAC and Remifentanil at a rate of 0.05-0.3 mcg/kg/min will be used. If additional hypotensive agents are required, an infusion of Esmolol at a rate of 25-200 mcg/kg/min will be initiated.
  Arms: Group Low
Other: Group Middle — In order to maintain arterial blood pressure within the range of 58-65 mmHg, Sevoflurane at a concentration of 0.5-1 MAC and Remifentanil at a rate of 0.05-0.3 mcg/kg/min will be used. If additional hypotensive agents are required, an infusion of Esmolol at a rate of 25-200 mcg/kg/min will be initiated.
  Arms: Group Middle

SUMMARY:
Controlled hypotension application is a commonly preferred anesthesia practice during surgical procedures, particularly in regions with rich tissue perfusion, aiming to reduce bleeding, enhance surgical field visibility, and mitigate potential complications. Preserving blood flow, especially to the brain, heart, and kidneys, is vital during this method. Previous studies on the subject have primarily focused on short-term effects regarding cognitive impairments, with limited research on the long-term impacts.

In our study, we aim to investigate how controlled hypotension application, administered to patients undergoing rhinoplasty or septoplasty surgery, specifically affects cerebral blood flow and its potential consequences on the development of short-term/medium-term/long-term cognitive impairments or delirium in the postoperative period.

DETAILED DESCRIPTION:
Nasal congestion is a health issue that affects approximately 70% of the general population, with nasal septal deviations being the most common cause . Various nasal septal surgeries, such as septoplasty or rhinoplasty, are performed to address aesthetic concerns related to curvature and correct deviations. The most common issue encountered during these operations is bleeding, which hinders the visibility of the surgical field. To prevent bleeding in the surgical area, the Trendelenburg position and controlled hypotension practices are frequently preferred . Controlled hypotension is defined as the intentional, elective, and controlled reduction of systolic blood pressure to 80-90 mmHg, the reduction of mean arterial pressure (MAP) to 50-65 mmHg, or a 30-50% reduction in baseline MAP.

Controlled hypotension is employed to shorten the duration of surgical procedures, reduce bleeding, decrease the need for blood transfusion, and enhance the quality of surgery by providing a satisfactory and clear surgical field without causing organ dysfunction.

Cognitive function is a mental process encompassing an individual's learning, understanding of oneself and the world, and acquired knowledge and beliefs about the surroundings. It covers higher brain functions such as consciousness, attention, learning, memory, perception, orientation, intelligence, action, emotion, imagination, problem-solving, decision-making, speech, reading, writing, and calculation. Cognitive function disorders are classified into delirium, dementia, amnestic disorder, cognitive disorder not otherwise specified, and postoperative cognitive dysfunction (POCD). POCD is a cognitive impairment that most commonly manifests with memory and concentration disturbances, diagnosable through neuropsychiatric tests. It is objectively measured cognitive decline beyond the expected duration for normal recovery from the physiological and pharmacological effects of anesthesia and surgery. POCD can persist from one day to years after surgery, increasing hospital stay and costs, affecting patients of all age groups, but more prevalent in older individuals. Early risk factors for POCD include anesthesia duration, low educational level, multiple surgical histories, postoperative infection, and respiratory complications. Late POCD, on the other hand, is only correlated with age among the identified risk factors. Bispectral index (BIS) and near-infrared spectroscopy (NIRS) monitoring are utilized in the perioperative process to prevent POCD . Studies have shown that lower BIS values in patients are associated with less development of postoperative cognitive dysfunction . The results suggest that deep anesthesia may have a protective effect by reducing cerebral metabolism and blood flow. Cerebral oxygenation monitoring has also demonstrated potential usefulness in preventing the development of postoperative cognitive dysfunction. Methods used for detecting postoperative cognitive dysfunction include direct interviews, questionnaires, mental status assessment tests, and neuropsychological tests . The most commonly used test among these is the Mini-Mental State Examination (MMSE). The MMSE, developed by Folstein and colleagues in 1975, evaluates cognitive functions and covers questions related to time and place orientation, memory and recall, attention and calculation, orientation, language, and visual structuring. A modified Mini-Mental test is used for those with no education. Both tests have a maximum score of 30, with 0-9 indicating severe cognitive impairment, 10-19 moderate cognitive impairment, 20-26 mild cognitive impairment, and 27-30 normal cognitive function.

Delirium is characterized by the acute onset, fluctuating course, and features such as disruption of cognitive functions due to organic causes, changes in the sleep-wake cycle, and decreased attention and perception . It is more common in intensive care units and the postoperative period, with advanced age being a risk factor for delirium due to the use of multiple medications and physical limitations. Various systemic illnesses and conditions related to the central nervous system can lead to delirium.

"Delirium, as it exhibits fluctuation throughout the day, is not always easily recognizable, and since only a medical professional can apply DSM criteria, the diagnosis may be overlooked. Screening and diagnostic tools have been developed to be easily and quickly applied using DSM criteria, allowing not only physicians but also nurses and healthcare personnel to use them.

Several assessment tools have been developed to easily and quickly detect and evaluate delirium. The Confusion Assessment Method (CAM) is a screening tool consisting of four features: (a) acute onset and fluctuating mental status, (b) inattention, (c) disorganized thinking, and (d) altered levels of consciousness.

Delirium can be diagnosed, especially using features (a) and (b), although (c) or (d) can be selectively used. For the intensive care unit, the CAM for the intensive care unit is a two-minute version of the CAM that can be easily applied in the intensive care unit with an accuracy of over 93%. Qualified personnel with appropriate training can apply CAM with high sensitivity.

The Richmond Agitation-Sedation Scale (RASS) is a tool used to assess the level of sedation/agitation. The DSM-5 guide states that a level of significantly decreased arousal above the level of coma (acutely onset) should be considered delirium, making RASS considered useful in diagnosing delirium.

The Delirium Rating Scale-Revised-98 (DRS-R-98) is useful in assessing the presence and severity of delirium but takes more time to administer than CAM. DRS-R-98 includes a relatively broader range of symptoms, comprising 3 diagnostic items and 13 severity items (total score ranging from 0 to 46, with a higher score indicating more severe delirium). It is suggested that a severity score of 15 or higher may indicate dementia or other psychiatric disorders.

Preventing the development of delirium is a primary approach in treatment. Identifying the causes of delirium and correcting the underlying organic disorder is the first treatment option. Measures to prevent delirium include ensuring the patient remains active, using auxiliary devices such as hearing aids and glasses when the patient is awake, avoiding restraints, and regulating the sleep-wake cycle. Therefore, nursing care is crucial. The secondary approach is treatment aimed at shortening the duration and reducing the severity of delirium in patients who develop delirium . Delirium is a condition where the sensitivity of the brain is increased. Medications that have anticholinergic side effects and lower the confusion threshold should be avoided. Delirium tremens, which occurs due to alcohol withdrawal, is treated with benzodiazepine derivatives . Benzodiazepine derivatives should not be used in treatment except for benzodiazepine deficiency and delirium tremens. If the patient with delirium is highly agitated and restless, haloperidol can be used as a sedative due to its low anticholinergic effect. Olanzapine, risperidone, and aripiprazole are second-generation antipsychotics. The use of these drugs is safe in delirium.

ELIGIBILITY:
Inclusion Criteria:

* who will undergo rhinoplasty or septoplasty surgery
* between the ages of 18-65
* classified as ASA class I-II

Exclusion Criteria:

* Patients with hypertension
* Patients with diabetes mellitus
* Patients with significant cardiac disease
* Patients with vascular disease with lung, kidney, or liver parenchymal diseases
* Patients with a history of cerebrovascular events
* Patients with hypovolemia
* those for whom perioperative controlled hypotension is contraindicated (including emergency surgeries, patients with bleeding diathesis, and those with heart valve disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Post Operative Cognitive Dysfunction with Mini Mental Test | 24 hours
  The assessment of patients' postoperative cognitive function will be conducted initially 24 hours after the surgery, and subsequently on the 7th day and at the 3rd month.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University Faculty of Medicince, Çorum, Merkez, Turkey (Türkiye)